CLINICAL TRIAL: NCT06780059
Title: Effects of Radiotherapy on Recurrence and Survival in Borderline and Malignant Phyllodes Tumors After R0 Resection: a Propensity Score Analysis
Brief Title: Effects of Radiotherapy in Borderline and Malignant Phyllodes Tumors After R0 Resection
Status: Completed | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yan Nie, Principal Investigator, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSKY-2024-1127-01
Record Dates: First submitted 2025-01-10; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Radiotherapy, Adjuvant; Phyllodes Breast Tumor; Prognosis
MeSH Terms: conditions — Phyllodes Tumor | interventions — Radiotherapy, Adjuvant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Phyllodes tumors patients who received radiotherapy afte R0 resection
  Interventions: Radiation: Adjuvant Radiotherapy; Procedure: R0 resection
- Phyllodes tumors patients who received R0 resection alone
  Interventions: Procedure: R0 resection

INTERVENTIONS:
Radiation: Adjuvant Radiotherapy — Postoperative Radiotherapy with 3D-CRT and IMRT Techniques Following R0 Resection in BoPT and MPT Patients
  Groups: Phyllodes tumors patients who received radiotherapy afte R0 resection
Procedure: R0 resection — Patients who received R0 resection (complete resection without tumor margin)

SUMMARY:
Breast phyllodes tumors (PT) are rare fibroepithelial neoplasms originating from stromal tissue and account for less than 1% of all breast tumors. The World Health Organization (WHO) classifies PT into benign, borderline, and malignant subtypes based on pathological features such as mitotic activity, cellular atypia, tumor margin invasion, and stromal composition 1. The presence of malignant heterologous elements characterizes the tumor as malignant 2. Surgery is the primary treatment. However, even after R0 resection, borderline phyllodes tumors (BoPT) and malignant phyllodes tumors (MPT) patients remain face a high risk of local recurrence, with rates of 15%-20% and 25%-30%, respectively. Moreover, metastases occur almost merely in MPT, with a distant metastasis rate reaching 22%.

Adjuvant radiotherapy has attracted attention for its potential to improve local control and reduce recurrence, but the role after R0 resection in PT patients remains unclear. Radiotherapy significantly reduces local recurrence rates in BoPT and MPT but shows no substantial benefit in benign cases. However, a meta-analysis by Yu et al. found that this effect is limited to MPT. Additionally, the effect of radiotherapy on survival rates in PT remains controversial. Most existing studies are retrospective and face limitations such as small sample sizes. The rarity of PT and conflicting evidence of impact of radiotherapy necessitate further study. While prospective trials are difficult due to limited cases, well-designed retrospective studies can offer valuable insights. In this study, the investigators also analyzed prognostic factors and identified subgroups to provide a clinical reference for the application of postoperative radiotherapy in BoPT and MPT patients.

ELIGIBILITY:
Inclusion Criteria:

* patients who were initially diagnosed with BoPT or MPT and underwent R0 resection surgery

Exclusion Criteria:

* patients who had their initial surgery at other hospitals without accurate baseline data
* patients who received radiotherapy before surgery
* those presenting with initial distant metastasis before treatment
* patients lost to follow-up after treatment
* patients with a history of or concurrent breast cancer or precancerous lesions in the ipsilateral breast or with breast cancer in the contralateral breast

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients pathologically diagnosed with BoPT and MPT who underwent surgery at three medical institutions in China: Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Sun Yat-sen University Cancer Center, and the Third Affiliated Hospital of Nanchang University.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-01-02 (Actual); Study Completion 2025-01-02 (Actual)

PRIMARY OUTCOMES:
5-year Local Recurrence-free Survival | Five years
  The time period from the initial R0 resection to either the detection of local recurrence or the final follow-up.

SECONDARY OUTCOMES:
5-year Overall Survival | Five years
  The time from the first R0 resection to either all-cause mortality or the last follow-up.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Third Hospital of Nanchang, Nanchang, Jiangxi

IPD SHARING:
Plan to Share IPD: No
no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Macdonald OK, Lee CM, Tward JD, Chappel CD, Gaffney DK. Malignant phyllodes tumor of the female breast: association of primary therapy with cause-specific survival from the Surveillance, Epidemiology, and End Results (SEER) program. Cancer. 2006 Nov 1;107(9):2127-33. doi: 10.1002/cncr.22228. PMID 16998937
- [Background] Pandey M, Mathew A, Kattoor J, Abraham EK, Mathew BS, Rajan B, Nair KM. Malignant phyllodes tumor. Breast J. 2001 Nov-Dec;7(6):411-6. doi: 10.1046/j.1524-4741.2001.07606.x. PMID 11843853
- [Background] Boutrus RR, Khair S, Abdelazim Y, Nasr S, Ibraheem MH, Farahat A, El Sebaie M. Phyllodes tumors of the breast: Adjuvant radiation therapy revisited. Breast. 2021 Aug;58:1-5. doi: 10.1016/j.breast.2021.03.013. Epub 2021 Apr 7. PMID 33865208
- [Background] Yu CY, Huang TW, Tam KW. Management of phyllodes tumor: A systematic review and meta-analysis of real-world evidence. Int J Surg. 2022 Nov;107:106969. doi: 10.1016/j.ijsu.2022.106969. Epub 2022 Oct 31. PMID 36328344
- [Background] Li J, Tsang JY, Chen C, Chan SK, Cheung SY, Wu C, Kwong A, Hu J, Hu H, Zhou D, Tse GM. Predicting Outcome in Mammary Phyllodes Tumors: Relevance of Clinicopathological Features. Ann Surg Oncol. 2019 Sep;26(9):2747-2758. doi: 10.1245/s10434-019-07445-1. Epub 2019 May 20. PMID 31111353
- [Background] Belkacemi Y, Bousquet G, Marsiglia H, Ray-Coquard I, Magne N, Malard Y, Lacroix M, Gutierrez C, Senkus E, Christie D, Drumea K, Lagneau E, Kadish SP, Scandolaro L, Azria D, Ozsahin M. Phyllodes tumor of the breast. Int J Radiat Oncol Biol Phys. 2008 Feb 1;70(2):492-500. doi: 10.1016/j.ijrobp.2007.06.059. Epub 2007 Oct 10. PMID 17931796
- [Background] Pezner RD, Schultheiss TE, Paz IB. Malignant phyllodes tumor of the breast: local control rates with surgery alone. Int J Radiat Oncol Biol Phys. 2008 Jul 1;71(3):710-3. doi: 10.1016/j.ijrobp.2007.10.051. Epub 2008 Jan 30. PMID 18234448
- [Background] Moffat CJ, Pinder SE, Dixon AR, Elston CW, Blamey RW, Ellis IO. Phyllodes tumours of the breast: a clinicopathological review of thirty-two cases. Histopathology. 1995 Sep;27(3):205-18. doi: 10.1111/j.1365-2559.1995.tb00212.x. PMID 8522284
- [Background] Md Nasir ND, Koh VCY, Cree IA, Ruiz BII, Del Aguila J, Armon S, Fox SB, Lakhani SR, Tan PH. Phyllodes tumour evidence gaps mapped from the 5th edition of the WHO classification of tumours of the breast. Histopathology. 2023 Apr;82(5):704-712. doi: 10.1111/his.14856. Epub 2023 Jan 30. PMID 36579383